CLINICAL TRIAL: NCT07226908
Title: Human Thalamus in Propagation of Temporal Lobe Seizures and Memory Formation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Josef Parvizi, Professor of Neurology and Neurological Sciences (Adult Neurology), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11354; 1R01NS137650-01A1 (NIH)
Record Dates: First submitted 2025-08-11; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy
Keywords: Intracranial Electroencephalography
MeSH Terms: conditions — Epilepsy | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epilepsy Patients with Thalamic Electrode Implants (Other): Patients will undergo cognitive testing and electrical stimulation experiments.
  Interventions: Other: Cognitive experiment; Other: Electrical stimulation of the brain

INTERVENTIONS:
Other: Cognitive experiment — Record brain activity during memory encoding
Other: Electrical stimulation of the brain — Measure accuracy and reaction time during cognitive tasks

SUMMARY:
The goal of the study is to examine how two key subregions of the human thalamus (ANT and PLV) are connected with other brain structures (Aim 1), how seizures involve the two thalamic subregions differently and how the map of cortico-thalamic ictal propagation matches the intrinsic connectivity maps identified in the same individuals (Aim 2), and the effect of ANT and PLV stimulations on memory formation (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* No medical or surgical contraindication to electrode implantation
* Patient capable of understanding the scope of our project or signing informed consent independently

Exclusion Criteria:

* Unable to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Cerebro-cerebral evoked potentials | During experiment up to 2 weeks
  To map thalamocortical and corticothalamic causal effective connectivity, the study team will use the well-known method of repeated single electrical pulse stimulation with intracranial EEG. Study team will measure the amplitude and timing to first peak of cerebro-cerebral evoked potentials (CCEPs).
fMRI BOLD activity | During experiment up to 2 weeks
  To map thalamocortical and corticothalamic functional connectivity, he study team will obtain 8 runs of 6mins resting state fMRIs. Study team will measure the correlation of BOLD activity across voxels of interest.
Epileptogenicity Index (EI) | During experiment up to 2 weeks
  The study team will identify seizure onset zones (SOZs) using the measure of Epileptogenicity Index (EI) applied to data collected through intracranial EEG, and will label the SOZs as medial temporal lobe epilepsy (mTLE) versus nonmedial TLEs.
Seizure propagation | During experiment up to 2 weeks
  Seizure propagation to ANT and PLV will be examined through intracranial EEG data within individuals by measuring EI and the propagation latencies from SOZ to ANT and PLV recording sites will be noted.
Coordinated activity across HPC and ANT | During experiment up to 2 weeks
  Successful memory encoding is associated with coordinated activity across hippocampus (HPC) and ANT (i.e., high frequency activity in ANT locked to the phase of hippocampal theta). Using intracranial EEG data, the study team will follow traditional analyses of changes in power in the canonical EEG bands (e.g., 3-7 Hz, theta band, 40-150 Hz, high gamma, etc.) as well as computationally derived aperiodic features of the signal [i.e., using the fitting oscillations & one over f (FOOOF) function]. Response onset latency of neural activity will determine with simultaneous recordings across HPC, ANT, and PLV how each ROI is engaged in time during a given experimental condition (i.e., encoding trials later recalled and trials not later recalled). We will also use validated methods of phase amplitude coupling (PAC) and intersite phase coherence (ISPC) to quantify cross regional relationships.
Cognitive task performance | During experiment up to 2 weeks
  In total, each patient will be asked to encode 200 words across the 5 sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Josef Parvizi, MD PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Once data collection and analysis for a Specific Aim is complete, we will share our data.
Supporting Information: Study Protocol
Time Frame: Within 2 years